CLINICAL TRIAL: NCT03463668
Title: Evaluation of the Efficacy of Duodenal Prostheses Not Covered Over 6 Years
Acronym: DYSPHAGIE
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: DYSPHAGIE-IPC 2017-036
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Digestive or Non-digestive Neoplasia Leading to Symptomatic Duodenal Stenosis
Keywords: duodenal stenosis; pyloric stenosis; digestive neoplasias; non-digestive neoplasias; duodenal prosthesis
MeSH Terms: conditions — Familial duodenal atresia; Pyloric Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- symptomatic non-covered duodenal prosthesis: Any symptomatic duodenal stenosis with symptomatic duodenal duodenal prosthesis between 2010 and 2017.
  Interventions: Device: uncovered metal duodenal prosthesis

INTERVENTIONS:
Device: uncovered metal duodenal prosthesis — Implantation of an uncovered metal duodenal prosthesis for symptomatic tumor stenosis

SUMMARY:
To assess the efficacy of duodenal prostheses for duodenal stenosis established for endoscopic pyloric or duodenal stenosis on dysphagia

DETAILED DESCRIPTION:
Duodenal prostheses have become, since the 2000s, the first-line treatment of unresectable duodenal tumoral stenosis. The technical success is greater than 90%, however the endoscopic revisions that are duodenal or biliary are frequent. The IPC as a center of interventional endoscopy is very often in charge of these stenoses. We wanted to evaluate the efficiency and the duration of this effectiveness in current situation. Is there still room for gastrojejunal gastrojejunal surgery or for the development of endoscopic gastrojejunal anastomoses?

ELIGIBILITY:
Inclusion Criteria:

* Any symptomatic duodenal stenosis with symptomatic duodenal duodenal prosthesis between 2010 and 2017.

Exclusion Criteria:

* Benign stenosis or covered metallic duodenal prosthesis (usually indicated for benign disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any symptomatic duodenal stenosis with symptomatic duodenal duodenal prosthesis between 2010 and 2017.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-22 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Dysphagia assessment | 7 years
  GOOSS = Gastric Outlet Obstruction Scoring System

SECONDARY OUTCOMES:
Rate of complications | 7 years
  Rate of complications
postoperative survival | 7 years
  defined as the time between the date of duodenal prosthesis insertion and the date of death or the latest news
Permeability duration of the duodenal stent | 7 years
  defined as the time between the date of the laying of the duodenal stent and date of patient's death or RED or surgery (exceptional case) or latest news
Rate of duodenal endoscopic resection at 1 and 3 months postoperatively | at 1 and 3 months postoperatively
  Rate of duodenal endoscopic resection at 1 and 3 months postoperatively
Rate of biliary endoscopic resection at 1 and 3 months postoperatively | at 1 and 3 months postoperatively
  Rate of biliary endoscopic resection at 1 and 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice CAILLOL, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiori E, Lamazza A, Volpino P, Burza A, Paparelli C, Cavallaro G, Schillaci A, Cangemi V. Palliative management of malignant antro-pyloric strictures. Gastroenterostomy vs. endoscopic stenting. A randomized prospective trial. Anticancer Res. 2004 Jan-Feb;24(1):269-71. PMID 15015607
- [Background] Johnsson E, Thune A, Liedman B. Palliation of malignant gastroduodenal obstruction with open surgical bypass or endoscopic stenting: clinical outcome and health economic evaluation. World J Surg. 2004 Aug;28(8):812-7. doi: 10.1007/s00268-004-7329-0. Epub 2004 Aug 3. PMID 15457364
- [Background] Jeurnink SM, Steyerberg EW, Hof Gv, van Eijck CH, Kuipers EJ, Siersema PD. Gastrojejunostomy versus stent placement in patients with malignant gastric outlet obstruction: a comparison in 95 patients. J Surg Oncol. 2007 Oct 1;96(5):389-96. doi: 10.1002/jso.20828. PMID 17474082
- [Background] ASGE guidelines enteral stents